CLINICAL TRIAL: NCT03562884
Title: Efficacy, Safety and Tolerability of a Split-dose of a New Bowel Cleansing Preparation (BLI800) in Adult Subjects Undergoing Colonoscopy: A Phase III, Multicentre, RANDOMIZED, 2 Parallel- Group, Comparative Versus Fortrans®, Non-inferiority, Investigator/Assessor-blinded Study
Brief Title: Efficacy, Safety and Tolerability of a New Bowel Cleansing Preparation (BLI800) in Adult Subjects Undergoing Colonoscopy
Acronym: EASY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: A-CN-58800-004
Record Dates: First submitted 2018-05-17; First posted 2018-06-20 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diagnosis Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLI800 (Experimental): BLI800 given orally as a split-dose: 1st dose the evening before colonoscopy (e.g. at 6:00 p.m.- 8:00 p.m.) and 2nd dose on the morning of colonoscopy, 10 to 12 hours after the evening dose (e.g. at 5:00 a.m.-7:00 a.m.)
  Interventions: Drug: BLI800
- Fortrans® (Active Comparator): Fortrans® given orally as a split dose: 1st dose the evening before colonoscopy (e.g. at 6:00 p.m - 8:00 p.m.) and 2nd dose on the morning of colonoscopy, 10 to 12 hours after the evening dose (e.g. at 5:00 a.m.-7:00 a.m.)
  Interventions: Drug: Fortrans®

INTERVENTIONS:
Drug: BLI800 — Two bottles of BLI800 are needed for appropriate cleansing of the bowel. Prior to administration, the content of each bottle must be diluted in water, using the cup provided, to a total volume of approximately 0.5 L, and must be followed by the ingestion of 1 additional litre of water.
  Arms: BLI800
Drug: Fortrans® — Fortrans® (Powder for Oral Solution) will be given according to Chinese approved Summary of Product Characteristics (SmPC). Fortrans® is provided as a powder for Polyethylene Glycol (PEG) based solution available in sachets containing a white powder readily miscible with water. The dosing for Fortrans® administration will be adapted to subjects' body weight as following: 1 L of solution for 15 to 20 kg, an average of 3 to 4 L (maximum 4 L).
  Arms: Fortrans®

SUMMARY:
The purpose is to demonstrate that BLI800 is non-inferior, on overall colon cleansing, to Fortrans® (a reference colonic lavage in China) administered in adult subjects scheduled to undergo a colonoscopy for a routinely accepted diagnostic indication.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent signed prior to any study related procedures.
* Male or female, at least 18 years old undergoing colonoscopy for a routine diagnostic indication, such as: a. Routine cancer screening b. Polyp or neoplasm history c. Diagnostic procedure for occult bleeding or anaemia d. Diarrhoea or constipation of unknown aetiology e. Inflammatory Bowel Disease (IBD) not in severe active phase
* In good clinical condition (physical exam and medical history)
* Adequate fluid balance, and adequate electrolyte balance (measured during screening K, Na, Cl, anion gap/bicarbonate/carbon dioxide content within normal/within ±10% of normal range)

Exclusion Criteria:

* Abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardise the subject's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.
* Advanced carcinoma or any other colon disease leading to excessive mucosal fragility.
* Known or suspected gastrointestinal (GI) obstruction, gastric retention, gastroparesis, or disorder of gastric emptying.
* Known or suspected ileus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-04-28 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with successful overall preparation based on a centrally assessed global BBPS score (for all segments) ≥ 6 (centralised assessment). | Through study completion, an average of 1 year
  Efficacy of BLI800 versus Fortrans® will be evaluated with the BBPS global score which ranges from 0 to 9. It will be blindly scored and evaluated by a centralised assessment (blinded assessors will assess the electronic record of colonoscopy and rate it).

SECONDARY OUTCOMES:
Assessment of cleanliness by investigators using the Boston Bowel Preparation Scale (BBPS) | Day 2
BBPS score by segment (0 to 3), scored in blind and evaluated by centralised assessment | Through study completion, an average of 1 year
Rate of polyp detection, evaluated by the investigator | Through study completion, an average of 1 year
Rate of adenomas detected, evaluated by the investigator | Through study completion, an average of 1 year
Rate of other lesions including cancer, evaluated by the investigator | Through study completion, an average of 1 year
Proportion of subjects for whom total colonoscopy could be completed, evaluated by the investigator | Through study completion, an average of 1 year
Investigator satisfaction evaluated by 5-point Likert scale score | Day 2
  Answers will be given on a 5-point rating scale.
Duration of the colonoscopy | Day 2
  Time from colonoscopy insertion to the time to reach the caecum.
Patient compliance with BLI800 versus Fortrans® | Through study completion, an average of 1 year
  The proportion of subjects who fully followed prescription will be analyzed. The compliance with the instructions of use provided in the prescription will be evaluated by the measurement of unused preparation and fluid intake recorded by the subject on the subject's leaflet. A subject will be considered as fully compliant with the instructions of use provided in the prescription if he drinks the whole preparation and any required further fluid intake.
Patient Satisfaction with BLI800 versus Fortrans® | Day 2
  Patient satisfaction will be evaluated by patient satisfaction scale. Satisfaction of bowel preparation will be performed by questionnaire assessing difficulty using bowel-cleansing preparations, ability to consume preparation, acceptability of taste, overall experience and questions regarding acceptance or refusal of future use of the same bowel preparation.
Patient tolerability with BLI800 versus Fortrans® | Day 2
  Evaluation of patient tolerability will be performed by patient tolerability questionnaire. Tolerability will be assessed by questionnaire recording the presence and intensity of specific symptoms (nausea, vomiting, abdominal pain, abdominal distension, and abdominal discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- China (10):
  - Peking University First Hospital, Beijing
  - Beijing Frendship hospital,Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - The Second Affiliated Hospital Zhe Jiang University of School, Hangzhou
  - Jiangsu Province Hospital, Nanjing
  - Zhong Shan Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan